CLINICAL TRIAL: NCT04179487
Title: The OPTICA Study - A Prospective Study Assessing the Quality and Safety of an Optimised CTPA Protocol in Pregnancy
Brief Title: The OPTICA Study - The Optimised Computed Tomography Pulmonary Angiography (CTPA) in Pregnancy, Quality and Safety Study
Acronym: OPTICA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College Dublin (Other)
Collaborators: Mater Misericordiae University Hospital (Other)
Responsible Party: Principal Investigator, Peter MacMahon, Professor Peter J Mac Mahon, MB BCH BAO, BMedSci, MRCPI, FFRRCSI., Mater Misericordiae University Hospital
Other Study IDs: 01
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Pulmonary Embolism; Pregnancy Related; Venous Thromboembolism
Keywords: pulmonary embolism; pregnancy; tomography xray computed; radiation dosage; negative predictive value
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant Patients with Suspected PE: Pregnant Patients with Suspected pulmonary embolism undergoing low dose CT pulmonary angiogram
  Interventions: Diagnostic Test: OPTICA CTPA Protocol

INTERVENTIONS:
Diagnostic Test: OPTICA CTPA Protocol — Low dose CT pulmonary angiogram protocol

SUMMARY:
A prospective multicentre study aiming to validate the clinical utility and safety of an optimised low-dose computed-tomography pulmonary angiogram (CTPA) protocol for suspected pulmonary embolism in pregnancy

DETAILED DESCRIPTION:
The OPTICA study is the first prospective study of a low-dose CTPA protocol for the pregnant population. It will define the achievable dose, image quality and safety of this protocol and provide an evidence base upon which modern CTPA protocols can be appropriately compared to scintigraphy for this population.

Pregnant women undergoing the specified low-dose CTPA protocol for suspected pulmonary embolism (PE), agreed across study sites with equivalent computed-tomography (CT) capabilities, will be included. Independent review of CTPAs by two radiology consultants, image data analysis and 3-month patient follow up will be performed.

The diagnostic algorithm employs chest-x-ray and lower limb Doppler if lower limb symptoms are present, followed by CTPA in cases where advanced imaging is required. D-dimer is permitted within the diagnostic algorithm for patients recruited after implementation of the updated 2019 "European Society of Cardiology guidelines for diagnosis and management of acute pulmonary embolism".

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant patients with a suspected pulmonary embolism
2. Age≥18 years

Exclusion Criteria:

1. Age < 18 years
2. Ultrasound proof of symptomatic proximal deep vein thrombosis
3. Contraindication to helical CT because of allergy to intravenous iodinated contrast or renal insufficiency (creatinine clearance <30 ml/min)
4. Treatment with full-dose therapeutic low molecular weight heparin or unfractionated heparin initiated 24 h or more prior to eligibility assessment
5. Treatment with vitamin K antagonists (coumarin derivates i.e. warfarin)
6. Unable or unwilling to consent
7. Unable to part-take in follow-up
8. Life expectancy <3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant Patients with Suspected pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 464 (Estimated)
Dates: Start 2018-05-29 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Venous Thrombo-Embolism (VTE) | 3 months
  3-month incidence of venous thromboembolism in pregnant patients in whom pulmonary embolism was excluded at baseline CT pulmonary angiogram.

SECONDARY OUTCOMES:
Maternal Effective Dose | 3 months
  Maternal Effective Dose
Breast Radiation Dose | 3 months
  Breast Dose
Foetal Radiation Dose | 3 months
  Foetal (Uterine) Dose
Signal to Noise Ratio | 3 months
  Image Quality - Objective Variable
Contrast to Noise Ratio | 3 months
  Image Quality - Objective Variable
Mean Pulmonary Trunk Enhancement | 3 months
  Image Quality - Objective Variable (Hounsfield Units)
Subjective Imaging Quality Grade | 3 months
  Subjective Imaging Quality Score: Score 1 - 5. Lowest score of 1 indicates a non diagnostic quality study. Best score of 5 indicates excellent quality / excellent opacification to the segmental pulmonary vessel level.

CONTACTS AND LOCATIONS:
Locations (1):
- Mater Misericordiae University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gillespie C, Foley S, Rowan M, Ewins K, NiAinle F, MacMahon P. The OPTICA study (Optimised Computed Tomography Pulmonary Angiography in Pregnancy Quality and Safety study): Rationale and design of a prospective trial assessing the quality and safety of an optimised CTPA protocol in pregnancy. Thromb Res. 2019 May;177:172-179. doi: 10.1016/j.thromres.2019.03.007. Epub 2019 Mar 13. PMID 30921536